CLINICAL TRIAL: NCT04803058
Title: A Safety and Tolerability Study of TCD601 (Siplizumab), a Human Anti-CD2 Antibody, Combined With Donor Bone Marrow Cell Infusion and Non-Myeloablative Conditioning, Including Fludarabine and Cyclophosphamide, for Tolerance Induction in Living Donor Renal Transplantation
Brief Title: A Study of TCD601 in the Induction of Tolerance in Renal Transplantation (PERSPECTIVE)
Acronym: PERSPECTIVE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ITB-Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD601A202
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): TCD601administered with non-myeloablative conditioning and standard of care immunosuppression
  Interventions: Biological: TCD601

INTERVENTIONS:
Biological: TCD601 — Investigational Product

SUMMARY:
The purpose of this study is to evaluate if TCD601 can induce allogeneic tolerance in living donor renal transplant recipients

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand the study requirements and provide written informed consent before any study assessment is performed
* Male or female patients ≥ 18 to 65 years of age
* Recipient of a renal transplant from a non-human leukocyte antigen (HLA)-identical but at least haploidentical, ABO compatible living donor

Key Exclusion Criteria:

* Women of child-bearing potential, unless willing to comply with the use of highly effective methods of contraception as defined by the protocol
* A history of cancer other than basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Recipient with anti-HLA donor-specific antibody (DSA)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
The safety, tolerability and activity of a Siplizumab-based conditioning regimen to induce renal allograft tolerance | 24 months
  The proportion of patients off immunosuppression with good safety and tolerability

SECONDARY OUTCOMES:
Incidence of biopsy proven acute rejection, death, and graft loss | 24 months
The incidence of DSA | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Killingsworth, Study Director — Nefro Avillion
Locations (3):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
- Samsung Medical University, Seoul, South Korea